CLINICAL TRIAL: NCT06941675
Title: Application of a Hybrid Closed-Loop Artificial Pancreas System in Patients With Latent Autoimmune Diabetes in Adults (LADA): An Open-Label, Randomized Controlled Trial
Brief Title: Hybrid Closed-Loop System in LADA Patients: A Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-2025-082
Record Dates: First submitted 2025-03-27; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Latent Autoimmune Diabetes in Adults (LADA)
MeSH Terms: conditions — Latent Autoimmune Diabetes in Adults

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Closed-Loop Artificial Pancreas System with CGM Group (Experimental): This group uses an open-source hybrid closed-loop artificial pancreas system with ultra-rapid-acting insulin (Novo Nordisk, Denmark). Daily insulin needs are calculated based on weight (0.3-0.6U/kg/day) & adjusted by the system. Physicians provide bolus instructions, entered by nurses. CGM & daily finger pricks are used for monitoring & calibration. The system predicts & prevents hypoglycemia, halting insulin when BG ≤ 4.4mmol/L. An alarm alerts for BG <3.9mmol/L.
  Interventions: Other: Hybrid Closed-Loop Artificial Pancreas System
- Conventional Insulin Pump Combined with CGM Group (Placebo Comparator): **According to the patient's weight, the total daily insulin requirement is calculated at a rate of 0.3 - 0.6 U/(kg·d) and distributed to pre-meal administrations based on the patient's specific condition. Blood glucose is monitored using a continuous glucose monitoring system in combination with daily fingerstick capillary blood glucose measurements (fasting blood glucose, and blood glucose 2 hours after breakfast, lunch, and dinner, for a total of 4 measurements). Insulin dosage is adjusted according to the patient's blood glucose levels until the blood glucose reaches the target level.**
  Interventions: Other: Hybrid Closed-Loop Artificial Pancreas System

INTERVENTIONS:
Other: Hybrid Closed-Loop Artificial Pancreas System — Hybrid Closed-Loop Artificial Pancreas System Group: Uses an open-source system with Novo Nordisk ultra-rapid-acting insulin (approval: J20050097, 3 mL: 300 U). Daily insulin dose calculated at 0.3-0.6 U/(kg*d) based on weight; system auto-adjusts basal rate. Physicians prescribe bolus doses, entered by nurses via AAPS software. Glucose correction uses CGM + 4 daily capillary tests (fasting, 2h post-meal). AAPS features hypoglycemia prediction suspend (pauses basal if glucose ≤4.4 mmol/L, resumes upon recovery) and alarms (<3.9 mmol/L, ensures nighttime alert).

SUMMARY:
Based on the difficulties in blood glucose control among the Latent Autoimmune Diabetes in Adults (LADA) population and the deficiencies of previous studies, this research aims to conduct a clinical comparative study. The short-term blood glucose control effects of the closed-loop system and the combination of a conventional insulin pump and Continuous Glucose Monitoring (CGM) in hospitalized LADA patients will be evaluated to explore the clinical application value of these methods in LADA patients. Moreover, this study aims to provide a more precise and personalized blood glucose management plan for LADA patients. As a slowly progressive subtype of autoimmune type 1 diabetes mellitus (T1DM), LADA patients have significant differences in pathological characteristics, clinical needs, and treatment effects compared with classical T1DM patients. However, they also face huge challenges in blood glucose management. This study will focus on LADA patients for the first time, especially the group of hospitalized patients, to fill the gap in this field. Meanwhile, by introducing the cutting-edge closed-loop system technology, it will provide new ideas and solutions for the clinical blood glucose management of LADA patients. Through a comparative analysis of the short-term blood glucose control effects of the closed-loop system and the combination of a conventional insulin pump and CGM, this study aims to provide more precise and personalized treatment strategies for LADA patients and promote the further development of diabetes treatment technologies.

DETAILED DESCRIPTION:
This study aims to compare the clinical effects of a hybrid closed-loop artificial pancreas system and a traditional insulin pump in hospitalized patients with Latent Autoimmune Diabetes in Adults (LADA) through a single-center, open-label, randomized controlled trial. Referring to the designs of similar clinical trials, the number of cases in each group of this study is determined to be 25, with a total of 50 cases. The study subjects are LADA patients hospitalized in the Department of Endocrinology of Shanxi Bethune Hospital from April 2025 to April 2027. The study design is as follows: Starting from the second 24-hour period after the patient's admission, with each subsequent 24-hour period as a monitoring unit, after collecting baseline data, the patients are randomly divided into two groups: the closed-loop system group and the control group. The closed-loop system group uses a hybrid closed-loop artificial pancreas system combined with Continuous Glucose Monitoring (CGM), while the control group continues to use a traditional insulin pump combined with CGM. During the study, both groups wear CGM devices for continuous monitoring, and relevant clinical data are collected during and after the treatment for statistical analysis to compare the short-term blood glucose control effects of the two intensive insulin treatment regimens in hospitalized LADA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old.
2. Meet the diagnostic criteria for LADA in the "Chinese Expert Consensus on the Diagnosis and Treatment of Latent Autoimmune Diabetes in Adults (2021 Edition)":

   * The onset age of diabetes is ≥ 18 years old.
   * Positive for islet autoantibodies or islet autoimmunity T cells.
   * Do not rely on insulin therapy for at least 6 months after the diagnosis of diabetes.
3. Patients are able to correctly use insulin pumps and CGM devices and have a certain learning ability and operational ability.
4. Baseline HbA1c > 7.0% or HbA1c > 6.0% combined with hypoglycemia.
5. Patients agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. The patient has been clearly diagnosed with type 2 diabetes or special types of diabetes.
2. The patient has experienced acute diabetic complications within the past 1 month, such as diabetic ketoacidosis, hyperglycemic hyperosmolar coma, etc.
3. The patient has severe symptoms of hypoglycemia intolerance.
4. The patient has skin diseases such as rashes and prurigo, or abnormal coagulation function.
5. The patient has diseases related to impaired glucose metabolism, such as uncontrolled hyperthyroidism, hypothyroidism, Cushing's syndrome, etc.
6. The patient has comorbid severe liver, kidney, gastrointestinal, hematological, brain, circulatory system diseases, etc.
7. The patient has other severe chronic diseases (such as malignant tumors, end-stage organ failure, etc.).
8. The patient has impaired consciousness or mental illness, lacks self-control, and cannot express clearly.
9. Lactating women, pregnant women, or women who plan to become pregnant during the trial period.
10. The patient is currently using or has used glucocorticoids or other drugs that interfere with glucose metabolism within 1 month before screening.
11. The patient is allergic to the drugs involved in the clinical diagnosis and treatment plan.
12. The patient is currently using other closed-loop systems.
13. People who are not suitable for conventional insulin pump treatment and those with contraindications.
14. The patient is known or suspected to have an insulin-allergic constitution and is allergic to adhesive tape, insulin pumps, or CGM devices.

Other situations where the researcher deems the patient unfit to participate in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Time required to achieve 70% TIR | 2 years
  Time in Range (TIR) refers to the percentage of time that blood glucose levels are within the target range of 3.9 to 10.0 mmol/L. The calculation formula is: TIR = (Time within the target range / Total time) × 100%
TIR achievement rate after 5 days of treatment | 5 days
  Time in Range (TIR) refers to the percentage of time that blood glucose levels are within the target range of 3.9 to 10.0 mmol/L. The calculation formula is: TIR = (Time within the target range / Total time) × 100%

SECONDARY OUTCOMES:
Blood Glucose Control Rate | 2 years
  The criteria for blood glucose target achievement are as follows: fasting blood glucose should be controlled within 4.0 - 7.0 mmol/L, postprandial blood glucose within 5.0 - 10.0 mmol/L, and blood glucose before going to bed within 4.4 - 7.8 mmol/L. The rate of blood glucose target achievement within 1 week of intensive insulin therapy will be statistically analyzed. The calculation formula is: Rate of blood glucose target achievement = (Number of patients achieving blood glucose targets / Total number of patients) × 100%
Time Below Range (TBR)、Time Above Range (TAR) | 2 years
  Time below the blood glucose target range, which is the percentage of time that blood glucose is below the target range of 3.9 mmol/L. The calculation formula is: TBR = (Time when blood glucose < 3.9 mmol/L in the target range / Total time) × 100%.
  Time above the blood glucose target range, which is the percentage of time that blood glucose is above the target range of 10.0 mmol/L. The calculation formula is: TAR = (Time when blood glucose > 10.0 mmol/L in the target range / Total time) × 100%.
Hypoglycemia Incidence Rate | 2 years
  The diagnostic criterion for hypoglycemia is a blood glucose level of 3.0 - 3.9 mmol/L. The hypoglycemia incidence rates during the treatment process in the two groups will be counted and compared. The diagnostic criterion for severe hypoglycemia is a blood glucose level < 3.0 mmol/L. The severe hypoglycemia incidence rates during the treatment process in the two groups will be counted and compared.
Inter-quartile Range (IQR) of Blood Glucose | 2 years
  The 25th and 75th percentile values of the blood glucose fluctuation range (inter - quartile range, IQR).
Average Daily Insulin Dosage | 2 years
  During the calculation period, record the specific dose of each injection every day.
Adverse Event | 2 years
  Count and compare the incidences of adverse events and serious adverse events during the treatment process between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
If there is a need to use data, please contact the person in charge and follow the relevant procedures to achieve data sharing. Without permission, do not use the data directly.